CLINICAL TRIAL: NCT05956184
Title: Intrauterine Device Insertion and Felt Pain: Which Method is Better?
Brief Title: Intrauterine Device Insertion and Felt Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Mohammad İbrahim Halilzade, Doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ACH-KHD-MIH-01
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Intrauterine Device Migration
Keywords: Pain; Intrauterine Devices; Conventional Technique; Direct Technique; IUD
MeSH Terms: conditions — Intrauterine Device Migration; Pain

STUDY DESIGN:
Intervention Model Description: Two groups as conventional method and direct method
Who Masked: Participant
Masking Description: The participants will not know which method would be applied to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convention Method Group (Active Comparator): Women who have an IUD inserted by conventional method will be asked to rate the most severe pain they experience during the procedure according to the Visual Analogue Scale (VAS) (from 0 to 10).
  Interventions: Device: Intrauterine Device Insertion
- Direct Method Group (Active Comparator): Women who have an IUD inserted by direct method will be asked to rate the most severe pain they experience during the procedure according to the Visual Analogue Scale (VAS) (from 0 to 10).
  Interventions: Device: Intrauterine Device Insertion

INTERVENTIONS:
Device: Intrauterine Device Insertion — All womens will be placed in a gynecological position and underwent a bimanual examination to better determine whether the uterus was in the anteverted or retroverted position. Subsequently, a speculum will be inserted, and the cervix will be disinfected with betadine. In the conventional method: the anterior lip of the cervix is grasped and pulled with Pozzi forceps, and after entering the uterine cavity with a hysterometry the IUD is inserted. In the direct method: the anterior lip of the cervix is grasped and pulled with Pozzi forceps, and without using hysterometry the IUD is directly inserted. The strings will be cut approximately 2-3 cm after the cervix, and the Pozzi forceps and speculum will be removed. The accuracy of the IUD placement will be confirmed using pelvic ultrasound. The process will take about five minutes.

SUMMARY:
The aim of this study is to compare the pain score between the direct method and the conventional method in patients who have undergone copper or hormonal intrauterine devices (IUD) for contraception and to find an answer to the question of which method is better.

DETAILED DESCRIPTION:
The intrauterine device (IUD) is one of the commonly used methods of contraception due to its effectiveness in providing reliable contraception, its ease of application, non-obstruction of sexual life, affordability, minimal absolute contraindications, and reversibility. Despite this increasing preference, concerns regarding the use of both levonorgestrel-releasing and copper IUDs due to the potential pain and fear of pain during insertion, which has hindered the adoption of this method.

Although the conventional method is used for intrauterine device insertion, the authors defined the direct method, also known as the torpedo technique, in 2006. IUD practitioners have started to prefer this direct method because it is simpler, faster and has fewer insertion steps than the conventional technique. However, IUD practitioners should apply the most painless and tolerable method to women who choose an IUD for contraception. Therefore, in order to understand which method is less painful, patients will be divided into 2 groups as those who have IUD inserted with the conventional method and those who have IUD inserted with the direct method. At the end of the procedure, participants in both groups will be asked to rate the most severe pain they experienced during the procedure according to the Visual Analogue Scale (VAS) (from 0 to 10).

In the conventional method: the anterior lip of the cervix was grasped and pulled with Pozzi forceps, and after entering the uterine cavity with a hysterometry the IUD was inserted.

In the direct method: the anterior lip of the cervix was grasped and pulled with Pozzi forceps, and without using hysterometry the IUD was directly inserted.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Preferring an intrauterine device for the contraceptive method

Exclusion Criteria:

* Patients with uterine leiomyoma
* Patients with endometriosis
* Patients with chronic pelvic pain
* Patients with familial mediterranean fever
* Patients who experienced complications during the procedure
* Patients who developed vasovagal reactions
* Patients who had previously used an IUD for any reason
* Patients with uterine anomalies

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women using an intrauterine device as a birth control method
Enrollment: 128 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Thirty minutes
  This is a numeric pain score evaluated as "painless" (score=0) and "worst pain" (score=10). Score <3 mild pain, 3-6 mild-moderate pain, and >6 moderate-to-severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad I Halilzade, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halilzade MI, Halilzade I, Turgay B, Kilickiran H, Turkmen O, Ozaksit MG. Effect of uterine sound on pain perception during intrauterine device insertion: A randomized trial. Medicine (Baltimore). 2025 Aug 1;104(31):e43721. doi: 10.1097/MD.0000000000043721. PMID 40760565